CLINICAL TRIAL: NCT04914897
Title: A Phase 2 Non-randomized, Open-label, Multi-cohort, Multi-center Study Assessing the Clinical Benefit of SAR444245 (THOR-707) Combined With Other Anticancer Therapies for the Treatment of Participants With Lung Cancer or Pleural Mesothelioma
Brief Title: A Study of SAR444245 Combined With Other Anticancer Therapies for the Treatment of Participants With Lung Cancer or Mesothelioma (Pegathor Lung 202)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16849; U1111-1254-0107 (Registry Identifier: ICTRP); MK-3475-B71 (Other: Merck Sharp & Dohme LLC.); KEYNOTE-B71 (Other: Merck Sharp & Dohme LLC.); 2020-005331-78 (EudraCT Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pleural Mesothelioma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy (Experimental): Participants with previously untreated Stage IV non-small cell lung cancer (NSCLC) and programmed cell death-ligand 1 (PD-L1) tumor proportion score (TPS) of >=50% were included in this cohort. Participants received pegenzileukin 24 microgram per kilogram (μg/kg) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion over 30 minutes every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as first-line [1L] therapy), until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort A2: NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy (Experimental): Participants with previously untreated Stage IV NSCLC and PD-L1 TPS of 1%-49% were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy (Experimental): Participants with NSCLC for whom standard of care (SOC) was not in their best interest or where no SOC was established were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as second-line or third-line [2/3L] therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort C1: Mesothelioma: Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy (Experimental): Participants with mesothelioma who had no SOC established and had experienced PD during or after at least one but no more than 2 prior regimens were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab

INTERVENTIONS:
Drug: THOR-707 — Intravenous infusion: solution for infusion
  Other Names: Pegenzileukin
Drug: Pembrolizumab — Intravenous infusion: solution for infusion
  Other Names: KEYTRUDA® or generic

SUMMARY:
The Primary Objective was:

-To determine the antitumor activity of SAR444245 in combination with other anticancer therapies.

The Secondary Objectives were:

* To confirm the dose and to assess the safety profile of SAR444245 when combined with other anticancer therapies.
* To assess other indicators of antitumor activity.
* To assess the pharmacokinetic (PK) profile of SAR444245 when given in combination with pembrolizumab.
* To assess the immunogenicity of SAR444245.

DETAILED DESCRIPTION:
The duration of the study for an individual participant started from the signature of the main informed consent and included a screening period of up to 28 days, a treatment period [max 35 cycles {cohorts A1, A2, and B1} = 735 days or until PD {cohort C1}], an end-of-treatment visit at least 30 days following the last administration of study drug (or until the participant receives another anticancer therapy, whichever is earlier), and a follow-up visit 3 months after treatment discontinuation and every 3 months following, until disease progression, or initiation of another antitumor treatment, or death, whichever is earlier

ELIGIBILITY:
Inclusion Criteria:

* Participant must have been ≥18 years of age (or country's legal age of majority if >18 years), at the time of signing the informed consent.
* Histologically or cytologically confirmed diagnosis of Stage IV NSCLC (cohorts A1, A2, and B1), or unresectable malignant pleural mesothelioma (cohort C1).
* Cohort A1: PD-L1 expression TPS ≥ 50%
* Cohort A2: PD-L1 expression TPS 1 - 49%
* Prior anticancer therapy
* Cohorts A1 and A2: No prior systemic therapy for advanced/metastatic NSCLC. Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the development of metastatic disease.
* Cohort B1: One prior anti-PD1/PD-L1 regimen (may include chemotherapy) plus one additional chemotherapy regimen
* Cohort C1: One or two prior systemic treatments that include pemetrexed-based regimen in combination with platinum agent.
* All cohorts must have had a measurable disease
* Mandatory baseline biopsy for the first 20 participants to enroll in cohorts A1, A2
* Cohort B1: Based on the Investigator's judgment, either docetaxel or pemetrexed is not the best treatment option for the participant.
* Females were eligible to participate if they were not pregnant or breastfeeding, not a woman of childbearing potential (WOCBP) or are a WOCBP that agrees:

  * to use approved contraception method and submit to regular pregnancy testing prior to treatment and for 150 days after discontinuing study treatment
  * to refrain from donating or cryopreserving eggs for 150 days after discontinuing study treatment.
* Males were eligible to participate if they agree to refrain from donating or cryopreserving sperm, and either abstain from heterosexual intercourse OR use approved contraception during study treatment and for at least 210 days after discontinuing study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria applied:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2.
* Poor bone marrow reserve
* Poor organ function
* Participants with baseline SpO2 ≤ 92%.
* Active brain metastases or leptomeningeal disease.
* History of allogenic tissue/solid organ transplant
* Last administration of prior antitumor therapy or any investigational treatment within 28 days or less than 5 times the half-life, whichever is shorter; major surgery or local intervention within 28 days.
* Has received prior IL-2-based anticancer treatment.
* Comorbidity requiring corticosteroid therapy
* Antibiotic use (excluding topical antibiotics) ≤14 days prior to first dose of IMP
* Severe or unstable cardiac condition within 6 months prior to starting study treatment
* Active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years
* Known second malignancy either progressing or requiring active treatment within the last 3 years
* Cohorts A1, A2, and C1: Prior treatment with an agent (approved or investigational) that blocks the PD1/PD-L1 pathway (participants who joined a study with an anti-PD1/PD-L1 but have written confirmation they were on control arm are allowed).
* Receipt of a live-virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (2):
  - Thomas Jefferson University Hospital Site Number : 8400009, Philadelphia, Pennsylvania
  - Thomas Jefferson University - North East Site Number : 8401009, Philadelphia, Pennsylvania
- Investigational Site Number : 0320002, CABA, Buenos Aires, Argentina
- Investigational Site Number : 0360002, Richmond, Victoria, Australia
- Chile (5):
  - Investigational Site Number : 1520005, Santaigo, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Temuco
- France (4):
  - Investigational Site Number : 2500006, Bordeaux
  - Investigational Site Number : 2500005, Paris
  - Investigational Site Number : 2500001, Saint-Herblain
  - Investigational Site Number : 2500003, Toulouse
- Italy (6):
  - Investigational Site Number : 3800005, Aviano (PN), Friuli Venezia Giulia
  - Investigational Site Number : 3800001, Rozzano, Milano
  - Investigational Site Number : 3800002, Orbassano, Torino
  - Investigational Site Number : 3800006, Bologna
  - Investigational Site Number : 3800004, Milan
  - Investigational Site Number : 3800008, Padua
- Investigational Site Number : 3920001, Sapporo, Hokkaido, Japan
- Poland (4):
  - Investigational Site Number : 6160002, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160003, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160004, Olsztyn, Warmian-Masurian Voivodeship
- South Korea (3):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Girona, Girona [Gerona]
  - Investigational Site Number : 7240004, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240001, Madrid
- Taiwan (3):
  - Investigational Site Number : 1580003, Taichung
  - Investigational Site Number : 1580002, Tainan
  - Investigational Site Number : 1580005, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16849 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25200&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 centers (corresponds to number of sites which screened at least one participant) in 11 countries. Out of 152 participants who were screened from 23 September 2021 to 07 October 2022, 106 participants were enrolled in the study and were assigned to 1 of the 4 cohorts (Cohorts A1, A2, B1, and C1) based on their disease type.
Pre-assignment Details: The study was terminated based on strategic sponsor decision not driven by any safety concerns. The Cohorts B2 and A3 were not initiated and no participants were enrolled.
  Note: Reason for not completed = Reason for permanent full intervention discontinuation.
Groups:
- Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy: Participants with previously untreated Stage IV non-small cell lung cancer (NSCLC) and programmed cell death-ligand 1 (PD-L1) tumor proportion score (TPS) of >=50% were included in this cohort. Participants received pegenzileukin 24 microgram per kilogram (μg/kg) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion over 30 minutes every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as first-line [1L] therapy), until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy: Participants with previously untreated Stage IV NSCLC and PD-L1 TPS of 1%-49% were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort C1:Mesothelioma: Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy: Participants with mesothelioma who had no SOC established and had experienced PD during or after at least one but no more than 2 prior regimens were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Period: Overall Study
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma: Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Started | 17 | 20 | 40 | 29
Completed | 5 | 1 | 1 | 0
Not Completed | 12 | 19 | 39 | 29
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1
Not completed — Poor compliance to protocol | 0 | 0 | 1 | 0
Not completed — Progressive disease | 5 | 14 | 30 | 21
Not completed — Adverse event: Not related to Coronavirus Disease 2019 (COVID-19) | 3 | 4 | 7 | 6
Not completed — Other | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The exposed population consisted of all participants who had given their informed consent and received at least one dose of study treatment (pegenzileukin or other anticancer therapies).
Groups:
- Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy: Participants with previously untreated Stage IV NSCLC and PD-L1 TPS of >=50% were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy: Participants with NSCLC for whom SOC was not in their best interest or where no SOC was established were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy: Participants with mesothelioma who had no SOC established and had experienced PD during or after at least one but no more than 2 prior regimens were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Total: Total of all reporting groups
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy | Total
Number analyzed (Participants) | 17 | 20 | 40 | 29 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.4) | 68.8 (8.4) | 63.6 (11.6) | 69.1 (10.7) | 66.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 13 | 8 | 35
  Male | 9 | 14 | 27 | 21 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 16 | 18 | 32 | 12 | 78
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 5 | 16 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cohorts A1 and A2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. CR. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 millimeter (mm) (<1 centimeter [cm]). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy
Number analyzed (Participants) | 17 | 20
percentage of participants | 41.2 [21.2 to 63.6] | 15.0 [4.2 to 34.4]

2. Primary Outcome: Cohorts B1: Objective Response Rate
Description: ORR was defined as the percentage of participants who had a confirmed CR or PR as per RECIST v1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 14 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 40
percentage of participants | 2.5 [0.1 to 11.3]

3. Primary Outcome: Cohorts C1: Objective Response Rate
Description: ORR was defined as the percentage of participants who had a confirmed CR or PR assessed by the investigator as per modified RECIST (mRECIST) v1.1. CR. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 29
percentage of participants | 3.4 [0.2 to 15.3]

4. Secondary Outcome: All Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened (according to the investigator's opinion) or became serious during the TE period.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment; approximately 28 months (Cohorts A1 and A2), 15 months (Cohort B1), and 25 months (Cohort C1)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 17 | 20 | 40 | 29
Participants
  TEAEs | 16 | 20 | 40 | 29
  TESAEs | 6 | 11 | 21 | 13

5. Secondary Outcome: All Cohorts: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Selected events that occurred during DLT observation period were considered as DLT unless due to PD or to a cause obviously unrelated to pegenzileukin. Selected events included: grade (G) 4 neutropenia for >=7 consecutive days, G3 or 4 neutropenia complicated by fever or microbiologically or radiographically documented infection, G3 or 4 thrombocytopenia associated with clinically significant bleeding that required clinical intervention; G3 or above alanine aminotransferase or aspartate aminotransferase in combination with a bilirubin >2 times upper limit of normal with no evidence of cholestasis or another cause such as viral infection or other drugs;G3 or above vascular leak syndrome, hypotension, and cytokine release syndrome;any other G3; G3 or 4 non-hematologic laboratory value; any death not clearly due to the underlying disease or extraneous causes;any toxicity that required permanent discontinuation of the study treatment(s).
Time Frame: From Day 1 to Day 21 of Cycle 1 (each cycle is 21 days)
Population: The DLT-evaluable population consisted of all exposed participants in the safety run-in who had been observed for at least 21 days. Any participants who had experienced a DLT during DLT observation period were also DLT-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 2 | 0 | 1 | 4
Participants | 0 | 0 | 1 | 0

6. Secondary Outcome: All Cohorts: Time to Response (TTR)
Description: TTR was defined as the time from the date of first study treatment administration to the first tumor assessment at which the overall response was recorded as PR or CR that was subsequently confirmed as per RECIST v 1.1 (NSCLC) and assessed by the investigator as per mRECIST v1.1 (mesothelioma). CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 27 months (Cohorts A1 and A2), 14 months (Cohort B1), and 24 months (Cohort C1)
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR or PR were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 7 | 3 | 1 | 1
months | 2.3 (0.8) | 3.4 (1.4) | 2.2 (NA) — NA indicates that the standard deviation (SD) was not estimable for 1 participant. | 4.1 (NA) — NA indicates that the SD was not estimable for 1 participant.

7. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: DOR was defined as time from date of first tumor assessment at which overall response was recorded as CR or PR that was subsequently confirmed to date of first documentation of objective PD before initiation of any post-treatment anti-cancer therapy or death due to any cause, whichever occurred first, as per RECIST v 1.1 (NSCLS) and assessed by investigator as per mRECIST v1.1 (mesothelioma). CR: disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. PD:at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this included baseline sum if that was smallest on study), in addition to relative increase of 20%, sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 7 | 3 | 1 | 1
months | NA [5.8 to NA] — NA indicates that the median and upper limit of 90% confidence interval (CI) were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that the median, lower limit, and upper limit of 90% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that the median, lower limit, and upper limit of 90% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that the median, lower limit, and upper limit of 90% CI were not estimable due to insufficient number of participants with events.

8. Secondary Outcome: All Cohorts: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants with clinical benefit: confirmed CR or PR as best overall response (BOR), or stable disease (SD) that lasted at least 6 months as per RECIST v 1.1 (NSCLS) and assessed by investigator as per mRECIST v1.1 (mesothelioma). CR: disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. BOR was the best response observed from start of the study treatment until PD, death, cut-off date or initiation of post-treatment anticancer therapy, whichever occurred first. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 17 | 20 | 40 | 29
percentage of participants | 58.8 [36.4 to 78.8] | 30.0 [14.0 to 50.8] | 5.0 [0.9 to 14.9] | 10.3 [2.9 to 24.6]

9. Secondary Outcome: All Cohorts: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the date of first study treatment to the date of the first documentation of objective PD, or death due to any cause, whichever occurred first as per RECIST v 1.1 (NSCLS) and assessed by investigator as per mRECIST v1.1 (mesothelioma). PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 17 | 20 | 40 | 29
months | 10.3 [4.2 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events. | 3.9 [2.1 to 8.7] | 2.1 [1.9 to 4.1] | 2.3 [2.1 to 4.0]

10. Secondary Outcome: All Cohorts: Plasma Concentrations of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of plasma concentrations of pegenzileukin. The pharmacokinetic (PK) parameters were calculated using non-compartmental method.
Time Frame: Days 2 and 3 of Cycle 1 (each cycle is 21 days)
Population: The PK population consisted of all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported. Limited or no participants returned on the Cycle 1 Day 3 for sample collection.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 15 | 17 | 25 | 22
nanogram/milliliter (ng/mL)
  Day 2 Cycle 1 | 214.7 (81.8) | 227.6 (77.7) | 212.0 (63.9) | 200.8 (61.4)
  Day 3 Cycle 1: number analyzed (Participants) | 2 | 0 | 1 | 4
  Day 3 Cycle 1 | 42.7 (14.8) |  | 121.0 (NA) — NA indicates that the SD was not estimable for 1 participant. | 56.3 (12.7)

11. Secondary Outcome: All Cohorts: Concentration at End of Infusion (Ceoi) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Ceoi of pegenzileukin.
Time Frame: Cycles 1, 2, 4, 7, 10, and 15 (each cycle is 21 days)
Population: The PK population consisted of all participants from exposed population with at least 1 PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported. Eventually, the participants discontinued as they progressed in the study. Hence, fewer participants at each cycle and no participants returned on Cycle 15 in Cohort B1 Arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 15 | 15 | 33 | 27
ng/mL
  Cycle 1 | 510.2 (164.1) | 434.1 (232.2) | 535.8 (402.6) | 457.0 (140.9)
  Cycle 2: number analyzed (Participants) | 13 | 15 | 28 | 20
  Cycle 2 | 445.8 (90.6) | 418.7 (215.3) | 585.6 (496.9) | 442.0 (131.7)
  Cycle 4: number analyzed (Participants) | 6 | 9 | 13 | 12
  Cycle 4 | 403.7 (122.6) | 413.9 (103.9) | 507.1 (168.6) | 400.4 (125.8)
  Cycle 7: number analyzed (Participants) | 7 | 3 | 7 | 6
  Cycle 7 | 509.3 (103.9) | 554.3 (129.3) | 590.3 (234.0) | 486.5 (251.3)
  Cycle 10: number analyzed (Participants) | 4 | 1 | 1 | 5
  Cycle 10 | 412.5 (109.4) | 483.0 (NA) — NA indicates that the SD was not estimable for 1 participant. | 152.0 (NA) — NA indicates that the SD was not estimable for 1 participant. | 443.0 (169.0)
  Cycle 15: number analyzed (Participants) | 1 | 1 | 0 | 1
  Cycle 15 | 352.0 (NA) — NA indicates that the SD was not estimable for 1 participant. | 265.0 (NA) — NA indicates that the SD was not estimable for 1 participant. |  | 567.0 (NA) — NA indicates that the SD was not estimable for 1 participant.

12. Secondary Outcome: All Cohorts: Number of Participants With Anti-Drug Antibodies (ADAs) Against Pegenzileukin
Description: Blood samples were collected at specified timepoints to assess the presence of ADAs against pegenzileukin. Treatment-emergent ADA was defined as at least one treatment-induced or treatment-boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA is presented.
Time Frame: as for outcome 4
Population: The ADA population consisted of all participants from the exposed population with at least one ADA result (positive, negative or inconclusive) after the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 13 | 9 | 18 | 8
Participants | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment; approximately 28 months (Cohorts A1 and A2), 15 months (Cohort B1), and 25 months (Cohort C1). All-cause mortality (death) was assessed from first dose of study treatment (Day 1) up to end of follow-up for death for each participant, approximately 32 months.
Description: Analysis was performed on the exposed population.
Groups:
- Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy: Participants with mesothelioma who had no SOC established were included in this cohort. Participants received pegenzileukin 24 μg/kg along with pembrolizumab 200 mg via IV infusion over 30 minutes q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Arm/Group | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy
All-Cause Mortality (participants affected / at risk) | 3/17 | 13/20 | 26/40 | 18/29
Serious Adverse Events (participants affected / at risk) | 6/17 | 11/20 | 21/40 | 13/29
Other Adverse Events (participants affected / at risk) | 16/17 | 18/20 | 38/40 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy (N=17) | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy (N=20) | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy (N=40) | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy (N=29)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 3 (4) | 7 (11) | 3 (3)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-Mediated Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillary Leak Syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal Oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1:NSCLC, PD-L1 TPS >=50%:Pegenzileukin 24 μg/kg + Pembrolizumab as 1L Therapy (N=17) | Cohort A2:NSCLC, PD-L1 TPS 1%-49%:Pegenzileukin 24 μg/kg+Pembrolizumab as 1L Therapy (N=20) | Cohort B1: NSCLC:Pegenzileukin 24 μg/kg+Pembrolizumab as 2/3L Therapy (N=40) | Cohort C1:Mesothelioma:Pegenzileukin 24 μg /kg+Pembrolizumab as 2/3L Therapy (N=29)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 5 (5) | 1 (1) | 7 (7) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular Device Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 1 (1) | 3 (3) | 4 (10) | 3 (7)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Immune-Mediated Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 6 (6) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1) | 5 (6)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sleep Deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital Oedema (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (5) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (10) | 2 (4) | 2 (2) | 4 (6)
Nausea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 6 (7) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1) | 5 (5) | 4 (7)
Hepatic Cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Immune-Mediated Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (3) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (7) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (7) | 4 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 6 (6)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sacral Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 7 (11) | 2 (2) | 13 (13) | 15 (17)
Chills (General disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (2) | 6 (7)
Feeling Hot (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Lithiasis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Amylase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood Magnesium Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Weight Decreased (Investigations) | 1 (1) | 1 (2) | 3 (3) | 2 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 10 (72) | 7 (45) | 19 (39) | 21 (75)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic sponsor decision not driven by any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04914897/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT04914897/SAP_001.pdf